CLINICAL TRIAL: NCT02181842
Title: Actos Tablets Specified Drug-use Survey <Survey on Glycemic Control in Type 2 Diabetic Patients With a History of Cerebral Infarction>
Brief Title: Pioglitazone Tablets Specified Drug-use Survey <Survey on Glycemic Control in Type 2 Diabetic Patients With a History of Cerebral Infarction>
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 237-019; JapicCTI-142568 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pioglitazone: Pioglitazone 15-30 mg, tablet, orally, once daily for up to 48 weeks before or after breakfast (the dose can be adjusted; however, the maximum daily dose should not exceed 45 mg).
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets
  Other Names: Actos Tablets

SUMMARY:
The purpose of this survey is to evaluate the effects on glycemic control and to evaluate the safety of long-term use of pioglitazone tablets (Actos Tablets) in type 2 diabetic patients with inadequate glycemic control and a prior history of cerebral infarction.

DETAILED DESCRIPTION:
This survey was designed to evaluate the effects on glycemic control and to evaluate the safety of long-term use of pioglitazone tablets (Actos Tablets) in type 2 diabetic patients with inadequate glycemic control and a prior history of cerebral infarction.

For adults, 15-30 mg of pioglitazone is usually administered orally once daily before or after breakfast. The dose should be adjusted depending on sex, age, and symptoms; however, the maximum daily dose should not exceed 45 mg.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with a prior history of cerebral infarction who meet all the following conditions, [1] to [3], at the time of enrollment in the survey:

  1. First onset of cerebral infarction was at least 24 weeks prior to enrollment
  2. HbA1c values ≥ 6.5% within 12 weeks prior to the start of treatment with Pioglitazone Tablets
  3. No prior history of treatment with Pioglitazone Tablets since the first onset of cerebral infarction

Exclusion Criteria:

* Patients who meet any of the following conditions, [1] to [5], shall be excluded from the survey:

  1. Contraindication for Actos Tablets
  2. Prior history of recurrence of cerebral infarction
  3. Prior history of cerebral hemorrhage or subarachnoid hemorrhage
  4. Complications or prior history of myocardial infarction, angina pectoris, cardiomyopathy, hypertensive heart disease, atrial fibrillation, atrial flutter, or valvular disease
  5. Reduced cardiac function (defined as an ejection fraction [EF] ≤ 40%)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2009-01-26 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 68 investigative sites in Japan, from 29 January 2009 to 30 June 2011.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with presence of cerebral infarction as medical history were enrolled to receive pioglitazone 15 milligram (mg) - 30 mg tablet, orally, once daily for up to 48 weeks.
Groups:
- Pioglitazone: Pioglitazone 15 mg - 30 mg, tablet, orally, once daily for up to 48 weeks before or after breakfast in participants based upon the disease severity. Participants will receive interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 246
Completed | 244
Not Completed | 2
Not completed — Case Report Forms Uncollected | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 163
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 244
Duration between Diagnosis of Cerebral Infarction and Start of Pioglitazone Therapy [Mean (Standard Deviation); unit: Days] — Duration between the first time of diagnosis of cerebral infarction and the start of Pioglitazone therapy was reported.
  Days | 1544.8 (1539.58)
Duration of Impaired Glucose Tolerance (IGT) [Count of Participants; unit: Participants] — Mean duration between start of study and first time of diagnosis of Impaired Glucose Tolerance (IGT) was reported.
  Participants
    < 1 year | 32
    1 - < 5 years | 63
    5 - < 10 years | 55
    ≥ 10 years | 60
    Unknown | 34
Predisposition to Hypersensitivity [Count of Participants; unit: Participants]
  Had no Predisposition to Hypersensitivity | 238
  Had Predisposition to Hypersensitivity | 5
  Unknown | 1
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 146
  Current Smoker | 43
  Ex-Smoker | 52
  Unknown | 3
Drinking Habits [Count of Participants; unit: Participants]
  Never Drank | 130
  Ex-Drinker | 44
  Current Drinker | 68
  Unknown | 2
Height [Mean (Standard Deviation); unit: centimete (cm)] | 159.43 (8.835)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 63.831 (10.9416)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 25.06 (3.399)
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had no Presence of Medical History | 176
    Had Presence of Medical History | 68
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had no Presence of Medical Complications | 12
    Had Presence of Medical Complications | 232
Initial Disease Type of Cerebral Infarction [Count of Participants; unit: Participants]
  Atherothrombotic Infarction | 99
  Lacunar Infarction | 129
  Cardioembolic Infarction | 6
  Other | 7
  Unknown | 3
Severity of Initial Cerebral Infarction [Count of Participants; unit: Participants]
  Small | 157
  Moderate | 52
  Multiple Small to Moderate-Sized | 31
  Severe | 3
  Unknown | 1
Modified Rankin Scale (mRS) at Start of Pioglitazone Therapy [Count of Participants; unit: Participants] — Modified Rankin Scale(mRS) is a scale for measuring the degree of disability or dependence in the daily activities and attributes the severity of cerebral infarction graded on a 7 point scale (0= No symptoms; 1= No significant disability; 2= Slight disability; 3= Moderate disability; 4= Moderately severe disability; 5= Severe disability; 6=Death). Higher scores indicate greater severity of neurological disability.
  Participants
    Grade 0 | 81
    Grade 1 | 103
    Grade 2 | 29
    Grade 3 | 17
    Grade 4 | 13
    Grade 5 | 0
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Good Glycemic Control (Reduction in Fasting Blood Glucose Level < 130 mg/dL)
Description: The reported data were percentage of participants who achieved good glycemic control at 48 Week. Good glycemic control was defined with fasting blood glucose level < 130 mg/dL.
Time Frame: 48 Week
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'Number of Participants Analyzed ' is number of participants analyzed at the given populations.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 116
Percentage of Participants | 42.2

2. Primary Outcome: Percentage of Participants Achieving Good Glycemic Control (Reduction in HbA1c Values < 6.9 %)
Description: The reported data were percentage of participants who achieved good glycemic control at 48 Week. Good glycemic control was defined with HbA1c (NGSP) Values < 6.9 %.
Time Frame: 48 Week
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here ' Number of Participants Analyzed ' is number of participants analyzed at the given populations.
Measure: Number; unit: Percent age of Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 115
Percent age of Participants | 40.0

3. Primary Outcome: Changes From Baseline in Laboratory Parameters (Systolic Blood Pressure (SBP)) at 48 Week
Description: Changes from baseline in laboratory parameter at 48 Week were reported. The reported data on this outcome measure is SBP as a one of laboratory parameters.
Time Frame: From Baseline, Up to 48 Week
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'Number of Participants Analyzed' is number of participants analyzed at the given populations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 117
mmHg | -6.9 (17.89)

4. Primary Outcome: Changes From Baseline in Laboratory Parameters (Diastolic Blood Pressure (DBP)) at 48 Week
Description: Changes from baseline in laboratory parameter at 48 Week were reported. The reported data on this outcome measure is DBP as a one of laboratory parameters.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 116
mmHg | -5 (11.96)

5. Primary Outcome: Changes From Baseline in Laboratory Parameters (High-Density Lipoprotein Cholesterol (HDL-Cholesterol)) at 48 Week
Description: Changes from baseline in laboratory parameter at 48 Week were reported. The reported data on this outcome measure is HDL-Cholesterol as a one of laboratory parameters.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 75
mg/dL | 3.97 (8.613)

6. Primary Outcome: Changes From Baseline in Laboratory Parameters (Low-Density Lipoprotein Cholesterol (LDL-Cholesterol)) at 48 Week
Description: Changes from baseline in laboratory parameter at 48 Week were reported. The reported data on this outcome measure is LDL-Cholesterol as a one of laboratory parameters.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 82
mg/dL | -1.85 (26.076)

7. Primary Outcome: Changes From Baseline in Glycosylated Hemoglobin (HbA1c) at 48 Week in Participants Stratified by Dose of Pioglitazone
Description: The reported data were changes from baseline in laboratory parameter, that is HbA1c (National Glycohemoglobin Standardization Program Criteria; NGSP), at 48 Week in participants stratified by specific characteristics, mean daily dose of pioglitazone, at the time of enrollment. Mean daily dose of pioglitazone at the time of enrollment were categorized into <15 mg, 15 to <30 mg, 30 <45 mg and 45 mg ≤ as planned (Note; final categorized number of participants was 0 in 45 mg ≤ group).
Time Frame: From Baseline, Up to 48 Week
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'n' is number of participants analyzed at the given populations.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent HbA1c
  <15 mg: number analyzed (Participants) | 6
  <15 mg | -0.84 (1.59)
  15 to <30 mg: number analyzed (Participants) | 153
  15 to <30 mg | -0.73 (0.806)
  30 <45 mg: number analyzed (Participants) | 30
  30 <45 mg | -0.98 (0.68)

8. Primary Outcome: Changes From Baseline in HbA1c at 48 Week in Participants Stratified by Levels of HbA1c
Description: The reported data were changes from baseline in laboratory parameter, that is HbA1c (NGSP), at 48 Week in participants stratified by specific characteristics, Levels of HbA1c, at the time of enrollment. Levels of HbA1c at the time of enrollment were categorized into <6.2%, 6.2 to <6.9%, 6.9 <7.4%, 7.4 <8.4%, and 8.4% ≤ as planned (Note; final categorized number of participants was 0 in <6.2% and 6.2 to <6.9% group).
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent HbA1c
  6.9 <7.4%: number analyzed (Participants) | 58
  6.9 <7.4% | -0.36 (0.504)
  7.4 <8.4%: number analyzed (Participants) | 90
  7.4 <8.4% | -0.83 (0.657)
  8.4% ≤: number analyzed (Participants) | 41
  8.4% ≤ | -1.17 (1.194)

9. Primary Outcome: Changes From Baseline in HbA1c at 48 Week in Participants Stratified by Gender
Description: The reported data were changes from baseline in laboratory parameter, that is HbA1c (NGSP), at 48 Week in participants stratified by specific characteristics, Gender, at the time of enrollment. Gender was categorized into male and female.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent HbA1c
  Male: number analyzed (Participants) | 128
  Male | -0.59 (0.729)
  Female: number analyzed (Participants) | 61
  Female | -1.11 (0.911)

10. Primary Outcome: Changes From Baseline in HbA1c at 48 Week in Participants Stratified by Levels of BMI
Description: The reported data were changes from baseline in laboratory parameter, that is HbA1c (NGSP), at 48 Week in participants stratified by specific characteristics, Levels of BMI, at the time of enrollment. Levels of BMI at the time of enrollment were categorized into <18.5 kg/m^2, 18.5 to <25 kg/m^2, 25 <30 kg/m^2, and 30 kg/m^2 ≤.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent HbA1c
  <18.5 kg/m^2: number analyzed (Participants) | 2
  <18.5 kg/m^2 | -0.6 (0)
  18.5 to <25 kg/m^2: number analyzed (Participants) | 74
  18.5 to <25 kg/m^2 | -0.73 (0.85)
  25 <30 kg/m^2: number analyzed (Participants) | 68
  25 <30 kg/m^2 | -0.81 (0.776)
  30 kg/m^2 ≤: number analyzed (Participants) | 13
  30 kg/m^2 ≤ | -1.3 (0.972)

11. Primary Outcome: Changes From Baseline in HbA1c at 48 Week in Participants Stratified by Presence of Companion Anti-Diabetes Drugs
Description: The reported data were changes from baseline in laboratory parameter, that is HbA1c (NGSP), at 48 Week in participants stratified by specific characteristics, presence of companion anti-diabetes drugs, at the time of enrollment. Presence of companion anti-diabetes drugs at the time of enrollment were categorized into Had presence of companion anti-diabetes drugs and Had no presence of companion anti-diabetes drugs.
Time Frame: From Baseline, Up to 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent HbA1c
  Had no Presence of Companion Drugs: number analyzed (Participants) | 50
  Had no Presence of Companion Drugs | -0.68 (0.922)
  Had Presence of Companion Drugs: number analyzed (Participants) | 139
  Had Presence of Companion Drugs | -0.8 (0.8)

12. Primary Outcome: Blood Glucose-Related Laboratory Parameters (Fasting Blood Glucose Level) at Each Time Point
Description: Fasting blood glucose level at baseline and 48 Week were reported as one of blood glucose-related laboratory parameters.
Time Frame: Baseline and 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 185
mg/dL
  Baseline | 172.62 (54.016)
  48 Week: number analyzed (Participants) | 114
  48 Week | 147.32 (43.102)

13. Primary Outcome: Blood Glucose-Related Laboratory Parameters (HbA1c Values) at Each Time Point
Description: HbA1c (NGSP) values at baseline and 48 Week were reported as one of blood glucose-related laboratory parameters.
Time Frame: Baseline and 48 Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Pioglitazone
Number analyzed (Participants) | 189
Percent
  Baseline | 7.83 (0.836)
  48 Week: number analyzed (Participants) | 115
  48 Week | 7.09 (0.777)

14. Secondary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to 48 Weeks
Population: Safety Analysis Set; The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 244
Participants | 23

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 16/244
Other Adverse Events (participants affected / at risk) | 7/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=244)
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 3
Hydrocephalus (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=244)
Oedema peripheral (General disorders) | 3
Weight increased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.